CLINICAL TRIAL: NCT02992080
Title: Determination of Circulating miRNAs as Diagnostic Markers of Lung Disease in Cystic Fibrosis
Brief Title: Small Circulating RNA as Molecular Markers of Lung Disease in Cystic Fibrosis
Acronym: MIRDIAMUCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 9548
Record Dates: First submitted 2016-09-07; First posted 2016-12-14 (Estimated); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Cystic Fibrosis
Keywords: Patient with Cystic Fibrosis; Patient without Cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cystic fibrosis Patients (Other)
  Interventions: Other: miRNAs isolation from blood samples of patients and control
- Patients without fibrosis cystic (Other)
  Interventions: Other: miRNAs isolation from blood samples of patients and control
- Cystic fibrosis Patients (secondary use of samples) (Other)
  Interventions: Other: miRNAs isolation from blood samples of patients and control

INTERVENTIONS:
Other: miRNAs isolation from blood samples of patients and control — Blood sample collection in specific PAXGene tubes

SUMMARY:
The aim of our study is to assess miRNAs expression profiles in the circuling blood of patients with cystic fibrosis and highlight "signatures" that could reflect the pulmonary status of patients

DETAILED DESCRIPTION:
The objective of this project is to study the circulating miRNA profiles in 40 patients with cystic fibrosis (5 samples which are acquired through a secondary use) and 40 healthy individuals to assess whether these biomolecules could be used as markers of the pulmonary disease in cystic fifbosis. Moreover by comparing miRNAs expression level between Cystic fibrosis (CF) patients with severe (n=20) or moderate (n=20) pulmonary impairment, we want to assess whether some of these miRNAs may be used as markers for the severity of CF pulmonary disease. The identification of sensitive and early markers, from a non-invasive sampling could enable more effective and early treatment of CF patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Cystic fibrosis (CF) (MIM#219700) who are compound heterozygous or homozygous for CF causing mutations Healthy controls non -smokers and free pulmonary disease

Exclusion Criteria:

* Participation or within the exclusion period of other clinicals trials Patients carrying mutations of clinical varying consequences or non CF-causing mutations
* smokers

Ages: 12 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Comparison of miRNAs expression between Cystic Fibrosis (CF) patients and healthy controls | After blood collection: 2 years
  Compare the distributions of miRNAs expression in blood samples of CF patients and to healthy controls

SECONDARY OUTCOMES:
Assesment of miRNAs expression in Cystic Fibrosis Patients depending on the pulmonary status | After blood collection 2 years
  Compare the distributions of miRNAs expression in blood samples of CF patients with mild lung disease and CF patients with severe lung disease

CONTACTS AND LOCATIONS:
Overall Officials: Caroline RAYNAL, PharmD, PhD, Principal Investigator — Montpellier University Hospital (CHU Montpellier) Montpellier University
Locations (2):
- France (2):
  - Montpellier University Hospital, Montpellier
  - Necker Hospital, Paris

IPD SHARING:
Plan to Share IPD: No